CLINICAL TRIAL: NCT07107867
Title: The Effect of Breastfeeding Counseling Provided During Pregnancy on Postpartum Breastfeeding Self-Efficacy and Infant Feeding Attitudes
Brief Title: The Effect of Breastfeeding Counseling on Postpartum Breastfeeding Self-efficacy and Infant Feeding Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, NUR FİDAN VARLIK, PhD Student, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-35766460-799
Record Dates: First submitted 2025-07-04; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Breastfeeding Education; Breastfeeding Self-Efficacy; Breastfeeding Attitude
Keywords: breastfeeding; breastfeeding self-efficacy; infant feeding attitude,; breastfeeding counseling; nursing
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to the intervention or control group using the website www.randomizer.org. This study was designed as a single-blind randomized controlled trial.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): The researcher, who had received certified training in breastfeeding counseling, conducted face-to-face interviews during the pretest phase. Mothers were informed about the purpose and nature of the study. After obtaining consent, pre-test data were collected from the pregnant women, and their group assignment was determined through randomization.
  Interventions: Behavioral: breastfeding counseling
- Control Group (No Intervention): Mothers in the control group who agreed to participate received only the hospital's standard breastfeeding care, with no additional intervention.

INTERVENTIONS:
Behavioral: breastfeding counseling — Pregnant women assigned to the intervention group then participated in a breastfeeding counseling training program held at the gynecology and obstetrics unit of an university training and research hospital. The training sessions lasted 60 to 90 minutes and included small groups of 5 to 6 participants, based on recommendations from the literature. The training was delivered through a slide presentation, and participants received a printed training booklet beforehand. Visual aids, including a baby model and breast model, were also used to enhance understanding. The training content was developed in line with infant feeding guidelines from UNICEF, the Turkish Ministry of Health, and relevant literature.
  Arms: Education Group

SUMMARY:
This study was conducted to determine the effect of breastfeeding counseling given to primiparous pregnant women before birth on breastfeeding self-efficacy and infant feeding attitudes in the postpartum period.

Hypotheses of this study:

H11: There is a difference in postpartum breastfeeding self-efficacy between the intervention group that received prenatal breastfeeding counseling and the control group.

H10: There is no difference in postpartum breastfeeding self-efficacy between the intervention group that received prenatal breastfeeding counseling and the control group.

H21: There is a difference between the intervention group that received prenatal breastfeeding counseling and the control group in terms of postnatal infant feeding attitude.

H20: There is no difference between the intervention group that received prenatal breastfeeding counseling and the control group in terms of postnatal infant feeding attitude.

DETAILED DESCRIPTION:
Breast milk is a natural source of nutrition that provides everything an infant needs for healthy physical growth, brain development, and a strong immune system. Starting breastfeeding within the first hour after birth, continuing exclusively for the first six months, and maintaining it alongside safe and appropriate complementary foods for up to two years or longer is one of the most effective ways to support a child's health and survival. However, only 43% of newborns worldwide are breastfed within that first hour. The highest early breastfeeding rates are found in Eastern and Southern Africa (65%), while the lowest are in East Asia and the Pacific (32%). In Türkiye, 71% of infants begin breastfeeding within the first hour after birth.

Although breastfeeding is a natural and physiological process, it also needs to be learned and it is not always easy to sustain. Several factors can make breastfeeding more challenging. These include the mother's young age, limited maternity leave for working mothers, lack of support from family or a partner, mode of birth, insufficient knowledge about breastfeeding, limited access to prenatal care and health education, low milk supply, difficulties with latching, medical issues affecting either the mother or the baby, and discomfort or embarrassment about breastfeeding in public.

According to the literature, face-to-face support from healthcare professionals promotes breastfeeding among healthy mothers and full-term infants. A mother's decision to start and continue breastfeeding, along with her attitudes and efforts toward it, is closely linked to her level of self-efficacy.

Self-efficacy beliefs play a key role in shaping an individual's behavior, motivation, and actions. Bandura (1977) defines self-efficacy as a person's belief or confidence in their ability to plan and carry out the actions necessary to handle future situations. In breastfeeding, self-efficacy is a crucial factor. It influences whether a mother chooses to breastfeed, how much effort she puts into it, whether she continues despite initial challenges, and how actively she works to improve her breastfeeding skills.

Breastfeeding self-efficacy during the prenatal period plays a key role in shaping a mother's intention and readiness to breastfeed after birth. This study examined the impact of breastfeeding counseling provided to pregnant women during the prenatal period on their breastfeeding self-efficacy and infant feeding attitudes in the postpartum period.

Hypotheses of this study:

H11: There is a difference in postpartum breastfeeding self-efficacy between the intervention group that received prenatal breastfeeding counseling and the control group.

H10: There is no difference in postpartum breastfeeding self-efficacy between the intervention group that received prenatal breastfeeding counseling and the control group.

H21: There is a difference between the intervention group that received prenatal breastfeeding counseling and the control group in terms of postnatal infant feeding attitude.

H20: There is no difference between the intervention group that received prenatal breastfeeding counseling and the control group in terms of postnatal infant feeding attitude.

Study Design This study is a single-blind randomized controlled experimental study. Population and Sample of the Study The population of the study consisted of pregnant women who attended the outpatient clinics of the Gynecology and Obstetrics Department at Ordu Training and Research Hospital, located in the Black Sea Region of Türkiye. 138 primiparous pregnant women were included in the study. 69 women were included in the training group and 69 women were included in the control group.

Pregnant women who were 18 years of age or older, had at least primary school education, had given birth for the first time, were in their 27th week of pregnancy or later, had no chronic disease, had no communication barriers, and agreed to participate in the study were included in the study.

Women were excluded from the study if they had any medical condition that might prevent breastfeeding, multiple pregnancy, multiparity, diagnosed mental illness, or were unwilling to continue participating in the study.

The independent variables of the study were age, education level and number of children.

The dependent variables of the study were receiving education on breastfeeding, the Iowa Infant Feeding Attitude Scale score, and the Breastfeeding Self-Efficacy Scale score.

The Control variables included a range of sociodemographic and obstetric characteristics such as age, education level, employment status, income level, spouse's education level, spouse's employment status, gestational week, health problems during pregnancy, structural nipple issues, prior breastfeeding education, and having a person around supporting breastfeeding.

Data Collection Tools Data were collected using several tools: a personal information form covering the participants' sociodemographic characteristics, the Antenatal Breastfeeding Self-Efficacy Scale-Short Form, the Postnatal Breastfeeding Self-Efficacy Scale-Short Form, and the Iowa Infant Feeding Attitude Scale. Before the breastfeeding counseling intervention, pregnant women completed these forms and scales themselves through face-to-face interviews. In the postpartum period, the same tools were completed by the participants via face-to-face interviews, telephone calls, or email.

Ethical Considerations Permission to use the scales was obtained via email from the authors. Ethical approval was obtained from the Ordu University Clinical Research Ethics Committee. Institutional approval was received from the Ordu Provincial Health Directorate. All pregnant women gave written and verbal informed consent to participate in the study.

ELIGIBILITY:
Inclusion Criteria: Pregnant women who agree to participate in the study,

* Are over 18 years old,
* Have at least primary school education,
* Are primiparous,
* Are in the 27th or more weeks of pregnancy,
* Have no chronic disease,
* Have no communication barriers will be included in the study.

Exclusion Criteria: Pregnant women who had medical indications that would prevent breastfeeding,

* Those who had multiple pregnancies,
* Those who were multiparous,
* Those who had a mental illness,
* Those who did not want to continue the research process,
* Those who could not be reached during the follow-up process were excluded from the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy Scale-Short Form | Data were collected with the BSES-SF in the prenatal period (enrollment), postpartum first week, postpartum first month and postpartum second month in the training and control groups. The evaluation of the data was made after December 2021.
  Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF), developed by Dennis (2003) to measure a mother's confidence in her ability to breastfeed.14 Aluş Tokat et al. (2010) adapted the scale for Turkish culture.19 The scale consists of two sub-dimensions: "technical" and "personal thoughts." It uses a Likert-type format ranging from 1 to 5, where 1 means "I am never sure" and 5 means "I am always sure." Scores range from 14 to 70, with higher scores indicating greater breastfeeding self-efficacy. In this study, the scale was used to assess self-efficacy before the breastfeeding counseling intervention. The Turkish adaptation reported a Cronbach's alpha of 0.87.
The Iowa Infant Feeding Attitude Scale | Data were collected using IIFAS in the prenatal period (enrollment), postpartum first week, postpartum first month, and postpartum second month in the training and control groups. Data analysis was performed after December 2021.
  The Iowa Infant Feeding Attitude Scale (IIFAS) was created to assess women's attitudes toward breastfeeding and to predict breastfeeding duration and choice of infant feeding method. The Turkish adaptation was conducted by Ekşioğlu et al. (2016).21 The scale consists of 17 items rated on a 5-point Likert scale, from 1 (strongly disagree) to 5 (strongly agree). Nine items reflect positive attitudes toward breastfeeding, while eight items reflect positive attitudes toward formula feeding; the formula feeding items (items 1, 2, 4, 6, 8, 10, 11, 14, and 17) are reverse scored. Scores can range from 17 to 85.20 There is no cut-off score. In the Turkish adaptation, the Cronbach's alpha was 0.71.

CONTACTS AND LOCATIONS:
Overall Officials: Nülüfer ERBİL, Prof., Principal Investigator — Ordu University
Locations (1):
- Ordu Üniversitesi Eğitim Araştırma Hastanesi, Altinordu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin CR, Ling PR, Blackburn GL. Review of Infant Feeding: Key Features of Breast Milk and Infant Formula. Nutrients. 2016 May 11;8(5):279. doi: 10.3390/nu8050279. PMID 27187450